CLINICAL TRIAL: NCT00789958
Title: A Phase II Trial of Adjuvant Capecitabine/Gemcitabine Chemotherapy Followed By Concurrent Capecitabine and Radiotherapy in Extrahepatic Cholangiocarcinoma (EHCC)
Brief Title: S0809: Capecitabine, Gemcitabine, and RT in Patients w/Cholangiocarcinoma of the Gallbladder or Bile Duct
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0809; S0809 (Other: SWOG); U10CA032102 (NIH); NCI-2009-00801 (Other: NCI)
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2016-09-22 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer
Keywords: cholangiocarcinoma of the extrahepatic bile duct; cholangiocarcinoma of the gallbladder; localized extrahepatic bile duct cancer; localized gallbladder cancer; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer; metastatic extrahepatic bile duct cancer; metastatic gallbladder cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Capecitabine; Gemcitabine; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adjuvant Chemo+ Chemoradiotherapy (Experimental): Adjuvant Chemotherapy
  * Capecitabine, 1500 mg/m^2/day, PO, Every 12 hrs on Days 1-14 of each cycle
  * Gemcitabine hydrochloride, 1000 mg/m^2, IV, Days 1 & 8 of each cycle
  Chemoradiotherapy
  -Capecitabine, 1330 mg/m^2/day, PO, Every 12 hrs, 7 days per week beginning the first day of RT and finishing the last day of RT
  Radiation (RT):
  3-dimensional conformal radiation therapy - 4,500 cGy over 5 weeks (5 days/week) in 180 cGy/fraction + 900 cGy during week 1 in 180 cGy fractions.
  intensity-modulated radiation therapy: 4,500 cGy over 5 weeks (5 days/week) in 180 cGy/fraction + 5,250 cGy in 210 cGy/fraction for a total of 25 fractions.
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: capecitabine — Adjuvant chemotherapy: 1500 mg/m^2/day, PO, Every 12 hrs on Days 1-14 of each cycle
  Chemoradiotherapy: 1330 mg/m^2/day, PO, Every 12 hrs, 7 days per week beginning the first day of RT and finishing the last day of RT
  Other Names: Xeloda; NSC-712807
Drug: gemcitabine hydrochloride — 1000 mg/m^2, IV, Days 1 & 8 of each cycle
  Other Names: Gemzar; NSC-619927
Radiation: 3-dimensional conformal radiation therapy — 4,500 cGy over 5 weeks (5 days/week) in 180 cGy/fraction + 900 cGy during week 1 in 180 cGy fractions.
  Other Names: 3D radiotherapy
Radiation: intensity-modulated radiation therapy — 4,500 cGy over 5 weeks (5 days/week) in 180 cGy/fraction + 5,250 cGy in 210 cGy/fraction for a total of 25 fractions.
  Other Names: IMRT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving more than one drug (combination chemotherapy) together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine together with gemcitabine followed by capecitabine and radiation therapy works in treating patients with cholangiocarcinoma of the gallbladder or bile duct.

DETAILED DESCRIPTION:
OBJECTIVES:

* To estimate the stratum-specific (R0 and R1) and overall 2-year survival probabilities of patients with extrahepatic cholangiocarcinoma treated with adjuvant chemotherapy comprising capecitabine and gemcitabine hydrochloride, followed by capecitabine and radiotherapy. (R0 stratum closed as of 12-15-11)
* To estimate the 2-year stratum-specific and overall disease-free survival and local disease-free survival of patients treated with this regimen.
* To assess the frequency and severity of toxicity in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to margin of resection (negative [R0] vs microscopically positive [R1]). (R0 stratum closed as of 12-15-11)

* Adjuvant chemotherapy: Patients receive oral capecitabine every 12 hours on days 1-14 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Chemoradiotherapy: Beginning in week 13, patients receive oral capecitabine every 12 hours on days 1-7. Patients also undergo concurrent three-dimensional or intensity-modulated radiotherapy on days 1-5. Treatment repeats weekly for 5-6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed extrahepatic cholangiocarcinoma of the gallbladder or bile duct, meeting at least 1 of the following criteria:

  * Pathological T2-4 disease
  * Pathological N1 disease
  * Positive margins (any T or N )
* Must have undergone potentially curative radical resection with negative (R0) or microscopically positive (R1) margins within the past 56 days and recovered (R0 stratum closed as of 12-15-11)
* No distant metastatic disease as indicated by a CT scan or MRI of the chest, abdomen, and pelvis within the past 42 days

  * Positive resected regional lymph nodes allowed
* No ampullary cancer

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC > 1,500/μL
* Platelet count > 100,000/μL
* Serum creatinine < 1.5 mg/dL
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* SGOT or SGPT < 2.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to swallow enteral medications and no requirement for a feeding tube
* No intractable nausea or vomiting
* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, requirement for IV alimentation, prior surgical procedures affecting absorptions. or uncontrolled inflammatory GI disease (e.g., Crohn disease, ulcerative colitis)
* No uncontrolled intercurrent illness including but not limited to any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Myocardial infarction or cerebrovascular accident within the past 3 months
  * Uncontrolled diarrhea
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No prior malignancy except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer, or other cancer from which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy for this disease
* No prior upper abdominal radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Ben-Josef, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (251):
- United States (251):
  - Regional Medical Center, Anniston, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Solano Medical Center, Vallejo, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - St. Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center - Shawnee Mission, Shawnee Mission, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Memorial Sloan-Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Memorial Sloan-Kettering Cancer Center - Rockville Centre, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

REFERENCES:
- [Derived] Ben-Josef E, Guthrie KA, El-Khoueiry AB, Corless CL, Zalupski MM, Lowy AM, Thomas CR Jr, Alberts SR, Dawson LA, Micetich KC, Thomas MB, Siegel AB, Blanke CD. SWOG S0809: A Phase II Intergroup Trial of Adjuvant Capecitabine and Gemcitabine Followed by Radiotherapy and Concurrent Capecitabine in Extrahepatic Cholangiocarcinoma and Gallbladder Carcinoma. J Clin Oncol. 2015 Aug 20;33(24):2617-22. doi: 10.1200/JCO.2014.60.2219. Epub 2015 May 11. PMID 25964250

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjuvant Chemotherapy + Chemoradiotherapy: Adjuvant Chemotherapy:
  Capecitabine, 1500 mg/m^2/day, PO, Every 12 hrs on Days 1-14 of each cycle; Gemcitabine hydrochloride, 1000 mg/m^2, IV, Days 1 & 8 of each cycle.
  Chemoradiotherapy:
  Capecitabine, 1330 mg/m^2/day, PO, Every 12 hrs, 7 days per week beginning the first day of RT and finishing the last day of RT; Radiation (RT): 3-dimensional conformal radiation therapy - 4,500 cGy over 5 weeks (5 days/week) in 180 cGy/fraction + 900 cGy during week 1 in 180 cGy fractions; intensity-modulated radiation therapy: 4,500 cGy over 5 weeks (5 days/week) in 180 cGy/fraction + 5,250 cGy in 210 cGy/fraction for a total of 25 fractions.
Period: Overall Study
Arm/Group | Adjuvant Chemotherapy + Chemoradiotherapy
Started | 105
Eligible and Analyzable | 79
Completed | 68
Not Completed | 37
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — Progression | 3
Not completed — not protocol specified | 1
Not completed — Not eligible/not analyzable | 26

BASELINE CHARACTERISTICS:
Population: All eligible and analyzable patients that received protocol treatment.
Arm/Group | Adjuvant Chemotherapy + Chemoradiotherapy
Number analyzed (Participants) | 79
Age, Continuous [Median (Full Range); unit: years] | 62 [26 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 66
  More than one race | 0
  Unknown or Not Reported | 2
Margin of Resection [Number; unit: participants]
  Negative (R0) | 54
  Microscopically positive (R1) | 25

OUTCOME MEASURES:

1. Primary Outcome: Stratum-specific (R0 and R1) 2-year Overall Survival
Description: Time to death is calculated from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients that received protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Patients With Negative Margins of Resection (R0): Eligible and analyzable patients that received a resection with negative (R0) margins.
- Patients w/Microscopically Positive Margin of Resection (R1): Eligible and analyzable patients that received a resection with microscopically positive (R1) margins.
Arm/Group | Patients With Negative Margins of Resection (R0) | Patients w/Microscopically Positive Margin of Resection (R1)
Number analyzed (Participants) | 54 | 25
percentage of participants | 67 [52 to 78] | 60 [38 to 76]

2. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 5 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary.
Measure: Number; unit: Participants
Arm/Group | Adjuvant Chemotherapy + Chemoradiotherapy
Number analyzed (Participants) | 79
Participants
  Anorexia | 1
  Cardiac troponin I (cTnI) | 1
  Constipation | 1
  Dehydration | 1
  Diarrhea | 6
  Fatigue (asthenia, lethargy, malaise) | 4
  Febrile neutropenia | 1
  Hemoglobin | 1
  Hemorrhage, GI - Duodenum | 1
  Hemorrhage, GI - Lower GI NOS | 1
  Hypotension | 1
  Lung Infection w/normal ANC or Gr 1-2 neutrophils | 1
  Skin Infection w/normal ANC or Gr 1-2 neutrophils | 1
  Infection-Other (Specify) | 1
  Leukocytes (total WBC) | 5
  Lymphopenia | 6
  Mucositis/stomatitis (clinical exam) - Oral cavity | 2
  Neuropathy: sensory | 1
  Neutrophils/granulocytes (ANC/AGC) | 35
  Phosphate, serum-low (hypophosphatemia) | 1
  Platelets | 2
  Potassium, serum-low (hypokalemia) | 2
  Rash/desquamation | 1
  Rash: hand-foot skin reaction | 10
  Sodium, serum-low (hyponatremia) | 1
  Syncope (fainting) | 1
  Thrombosis/embolism (vascular access-related) | 1
  Thrombosis/thrombus/embolism | 1
  Ulcer, GI - Duodenum | 1
  Ventricular arrhythmia - Ventricular tachycardia | 1

3. Secondary Outcome: 2-year Overall Survival for All Patients
Description: as for outcome 1
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients that received protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adjuvant Chemotherapy + Chemoradiotherapy
Number analyzed (Participants) | 79
percentage of participants | 65 [53 to 74]

4. Secondary Outcome: 2-year Stratum-specific Disease-free Survival
Description: Disease-free survival is calculated from date of registration to date of first documentation of relapse or death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients that received protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Negative Margins of Resection (R0) | Patients w/Microscopically Positive Margin of Resection (R1)
Number analyzed (Participants) | 54 | 25
percentage of participants | 54 [40 to 66] | 48 [27 to 65]

5. Secondary Outcome: 2-year Disease-free Survival in All Patients
Description: as for outcome 4
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients that received protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adjuvant Chemotherapy + Chemoradiotherapy
Number analyzed (Participants) | 79
percentage of participants | 52 [40 to 62]

6. Secondary Outcome: 2-year Stratum-specific Local Relapse Rate
Description: Local relapse is any evidence of new disease within the primary tumor bed or the regional (retroperitoneal, celiac, and portal vein nodes) lymphatics (these areas are to be encompassed within the radiation fields).
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients that received protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Negative Margins of Resection (R0) | Patients w/Microscopically Positive Margin of Resection (R1)
Number analyzed (Participants) | 54 | 25
percentage of participants | 9 [2 to 17] | 16 [2 to 30]

7. Secondary Outcome: 2-year Overall Local Relapse Rate
Description: as for outcome 6
Time Frame: Up to 2 years from registration
Population: Eligible and analyzable patients that received protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adjuvant Chemotherapy + Chemoradiotherapy
Number analyzed (Participants) | 79
percentage of participants | 11 [4 to 18]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Eligible patients who received any treatment and were assessed for adverse events are included in the adverse event summaries.
Arm/Group | Adjuvant Chemotherapy + Chemoradiotherapy
Serious Adverse Events (participants affected / at risk) | 2/79
Other Adverse Events (participants affected / at risk) | 78/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Chemotherapy + Chemoradiotherapy (N=79)
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 1
Hemorrhage, GI - Duodenum (Gastrointestinal disorders) | 1
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 1
Thrombocytopenia (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Chemotherapy + Chemoradiotherapy (N=79)
Low hemoglobin level (Blood and lymphatic system disorders) | 45
Constipation (Gastrointestinal disorders) | 24
Diarrhea (Gastrointestinal disorders) | 35
Distention/bloating, abdominal (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 7
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 17
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 49
Pain - Abdomen NOS (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 15
Edema: limb (General disorders) | 11
Fatigue (asthenia, lethargy, malaise) (General disorders) | 64
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 17
Pain-Other (General disorders) | 11
Rigors/chills (General disorders) | 5
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 21
AST, SGOT (Investigations) | 22
Alkaline phosphatase (Investigations) | 21
Bilirubin (hyperbilirubinemia) (Investigations) | 6
Leukocytes (total WBC) (Investigations) | 42
Lymphopenia (Investigations) | 21
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 52
Platelets (Investigations) | 26
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 17
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 25
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 8
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6
Pain - Back (Musculoskeletal and connective tissue disorders) | 6
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 5
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 9
Neuropathy: sensory (Nervous system disorders) | 24
Pain - Head/headache (Nervous system disorders) | 12
Taste alteration (dysgeusia) (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 11
Mood alteration - anxiety (Psychiatric disorders) | 8
Mood alteration - depression (Psychiatric disorders) | 6
Urinary frequency/urgency (Renal and urinary disorders) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 9
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 7
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 27
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No